CLINICAL TRIAL: NCT00880035
Title: M.U.S.I.C (MUSicotherapy in the Intensive Care) Interventional, Pilot, Cross-Over, in Mechanically-Ventilated Patients on ICU Ward
Brief Title: Efficacy of Music on Reduction of Sedative Drugs in Mechanically Ventilated Intensive Care Unit Patients
Acronym: MUSIC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de Recherche Clinique CHUS (Unknown)
Responsible Party: Olivier Lesur (PI) (Catherine St-Pierre co-PI), CRC-CHUS
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08-105-R2; CRC-PAFI-09
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Sedative Drug Consumption; Mechanically Ventilated ICU Patients
Keywords: sedative drug; stress; music; mechanical ventilation; IL-6; cortisol; prolactin; CRP; copeptin
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A: day 1 = music, day 2 = washout, day 3 = headphone without music
  Interventions: Device: MP3 music program listening
- Group B (Experimental): Group B: day 1 = headphone without music, day 2 = washout, day 3 = music
  Interventions: Device: MP3 music program listening

INTERVENTIONS:
Device: MP3 music program listening — 3 days with two 1 hour periods of headset music listening (1 day on, 1 day wash-out, 1 day off)

SUMMARY:
Major objective: a three-days interventional cross-over trial [one day music on, one day wash-out, one day music off][two periods of listening/day], to evaluate:

1. Impact on sedative drug consumption.
2. Alteration of stress neuropeptide blood concentrations.

Population: mechanically-ventilated ICU patients

The investigators hypothesize the music will decrease the need of sedative drugs and reduce the concentration of neuropeptides in circulation.

DETAILED DESCRIPTION:
The study will imply patients mechanically ventilated for more than 3 days, that require sedation with benzodiazepine and narcotics.

There will be two groups both of exposed to music and placebo (headphones without music). The study will be simple blind.

Sedation scale will be followed regularly. Vitals signs and adjustment of sedation will be recorded by the nurse on the ward. Blood test will be taken before and after placement of headphones in the morning. We will measure IL-6, cortisol, copeptin, prolactin, CRP.

We will analyse the total reduction dose of sedation and analgesia on a daily basis. We will consider a fall of 20% of medication to be significative.

ELIGIBILITY:
Inclusion Criteria:

* adults older than 18 years old
* expected time of mechanical ventilation of more than 72 hours
* sedation needs for a scale of Sedation-Agitation Scale (SAS) more than 1

Exclusion Criteria:

* hearing impairment
* pregnancy
* needs of vasopressin
* needs of curarisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
sedative drug consumption in mechanically ventilated ICU patients | 3 days

SECONDARY OUTCOMES:
stress neuropeptide blood content evolution with MUSIC listening | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lesur, MD, Principal Investigator — CHUS and Université de Sherbrooke
Locations (1):
- CHUS, Sherbrooke, Quebec, Canada